CLINICAL TRIAL: NCT02716207
Title: Mono-Center Phase ǀ Study on Dose Escalation of Stereotactic Body Radiotherapy (SBRT) Treating Pancreatic Cancer Patients With CyberKnife
Brief Title: Phase ǀ Study on Pancreatic Cancer Treated by CyberKnife
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Director of Radiation Oncology Department, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChanghaiH001
Record Dates: First submitted 2016-01-06; First posted 2016-03-23 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Pancreatic Tumor
Keywords: Stereotactic Body Radiotherapy (SBRT); CyberKnife; Dose Escalation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Maximal tolerated dose with CyberKnife (Experimental): SBRT will be delivered in 5 fractions within 1 to 2 weeks by the following schedule: Doses of 7 Gy, 7.5 Gy, 8 Gy, 8.5 Gy, 9 Gy, 9.5 Gy x 5 with BED10 in correspondence to 59.5 Gy, 65.6 Gy, 72 Gy, 78.6 Gy, 85.5 Gy, 92.6 Gy respectively while meeting with normal tissue constraints. A minimum of three patients will be included for each dosage level. And an interval is four weeks between each dose level. In case patient presents III/IV GI toxicity, three additional patients will be included at the same dose level. The Maximal Tolerated Dose will be defined as the dose for which at least 2 patients in 3, or at least 3 patients in 9, will present with a limiting toxicity.
  Interventions: Device: CyberKnife

INTERVENTIONS:
Device: CyberKnife — Radiation Therapy

SUMMARY:
The maximum tolerated dose on locally advanced unresectable pancreatic tumor treated with CyberKnife SBRT will be evaluated.

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth-leading cause of cancer-related death in the world. It is characterized by metastatic spread and local failure and seldom detected in its earlier stages. For locally advanced stage pancreatic cancer, the complete surgical removal is hard to achieve.

Stereotactic body radiotherapy (SBRT) with CyberKnife for unresectable pancreatic tumor is a relatively new treatment option made available because of significant improvements in diagnostic imaging and radiation delivery techniques. Different from the conventional radiotherapy, radiation dose is delivered in fewer fractions and higher fractional doses in SBRT. Gurka (1) reported that 14 patients received SBRT with prescription dose of 25 Gy in five fractions with biologically equivalent doses (BED) of α/β=10 in correspondence to 37.5Gy. Grade 1 to 2 gastrointestinal toxicity (no grade 3 or 4 radiation-related toxicities) was observed two weeks after treatment. Two patients had a partial response, and 12 patients were with stable diseases. In the previous dose escalation study, a single fraction up to15 Gy, 20 Gy, 25 Gy which is an equivalent BED10 to 37.5 Gy, 60 Gy, 87.5 Gy respectively is recommended by Koong AC (2) and his team. Even though the local control rate is 100%, the follow up is short and the sample size of 15 patients is relatively small. Moreover, the late toxicity is not investigated. And with single fraction scheme, higher late gastrointestinal (GI) toxicities were reported (2,3,4). In the meanwhile, investigators (5, 6) from South Korea examined that a Dmax of 35Gy and 38Gy in 3 fractions (BED10 to 75.8Gy and 86.1Gy) of SBRT correlated with a 5% and 10% rate of grade 3 of gastroduodenal toxicity for abdominal malignant tumor, respectively.

Chuong (7) used 5 fractions to potentially decrease the risk of late normal tissue injury compared with 1 to 3 fractions commonly used in other institutions. Assuming α/β=3, the BED3 delivered to normal tissue in this study (using a mean 36.4 Gy in 5 fractions to the high dose PTV) was 125 Gy, which is lower than the mean BED3 from other series, the corresponding values from Boston and Stanford were 153.7 Gy (mean, 32.96 Gy in 3 fractions) and 233.3 Gy (mean, 25Gy in 1 fraction), respectively (8, 9). And a relatively lower incidence of grade ≥3 late adverse effects (5.3% VS 9%) was observed.

Since the treatment modality and dose are still under exploratory stage, we propose to conduct a Phase I study determining the maximum tolerated dose of CyberKnife SBRT on dose escalation for the treatment of locally advanced pancreatic tumor based on a 5 fractions treatment regimen. A prescription dose of 35-47.5 Gy in five fractions was chosen, with an equivalent to the traditional dose of 2 Gy in 25-39 fractions of BED10. And this is assumed to be the safe and effective dose for unresectable pancreatic cancer patients.

Study Procedure:

CyberKnife SBRT body fixation (vacuum-bag) will be used in immobilizing the body, the arms and the legs.

* Patients will undergo a plain CT as well as an enhanced pancreatic parenchymal CT for radiation treatment planning and target delineation.
* SBRT will be delivered on CyberKnife with Synchrony Respiratory Tracking system. The tumor will be tracked with implanted fiducial markers by Fiducial Tracking System. Treatment will be delivered in 5 fractions within 1 to 2 weeks at the discretion of the investigator.
* A body fixation (vacuum-bag) will be used in immobilizing the body, the arms (both arms are along the body) and the legs.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable pancreatic adenocarcinoma or unsuitable/unwilling for resection which is proved by biopsy.
* A life expectancy of >3months
* Eastern Cooperative Oncology Group (ECOG) status ≤2
* Tumor size < 5 cm
* Tumor location: Head of pancreas
* Patients must be able to undergo contrast enhanced CT for planning
* Absolute neutrophil count (ANC) ≥ 1.5 ×109 cells/L
* Leukocyte count≥ 3.5 ×109cells/L
* Platelets ≥ 70×109cells/L
* Hemoglobin ≥ 8.0 g/dl
* Albumin > 2.5 g/dL
* Total bilirubin < 3 mg/dL
* Creatinine < 2.0 mg/dL
* INR < 2 (0.9-1.1)
* Aspartate transaminase (AST) <2.5 × Upper Limit of Normal (ULN )(0-64U/L)
* Alanine aminotransferase (ALT) <2.5 × ULN(0-64U/L)
* Both men and women and members of all races and ethnic groups are eligible for this study
* Ability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document
* Tumor markers and lab test should be done less than 1 week before recruitment

Exclusion Criteria:

* Prior surgery, chemotherapy or radiation for the pancreatic tumor
* Prior radiotherapy to the upper abdomen, evidence of metastatic disease such as nodal or distant metastases by abdomen CT and chest CT or FDG PET-CT
* Contraindication to receiving radiotherapy
* Distance between gross tumor volume (GTV) (lesion) and luminal structures (including liver, stomach, duodenum, small or large bowel) is<5 mm
* Women who are pregnant
* Participation in another clinical treatment trial while on study
* Patients in whom fiducial implantation was not possible

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose will be determined | 2 years
  The maximal tolerated dose will be defined as the dose for which at least 2 patients in 3, or at least 3 patients in 9, will present with a limiting toxicity.

SECONDARY OUTCOMES:
The acute toxicities following SBRT will be determined. | 1 year
  The acute toxicities are determined by RTOG Acute Radiation Morbidity Scoring Criteria.
The late toxicities following SBRT will be determined. | 1 year
  The late toxicities are determined by RTOG/EORTC Late Radiation Morbidity
Pain intensity will be determined. | 1 year
  Pain intensity is assessed by the numeric rating scales 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Huo Jun Zhang, MD., PH.D, Principal Investigator — Changhai Hospital
Locations (2):
- China (2):
  - Huojun Zhang, Shanghai, Shanghai Municipality
  - HuojunZhang, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gurka MK, Collins SP, Slack R, Tse G, Charabaty A, Ley L, Berzcel L, Lei S, Suy S, Haddad N, Jha R, Johnson CD, Jackson P, Marshall JL, Pishvaian MJ. Stereotactic body radiation therapy with concurrent full-dose gemcitabine for locally advanced pancreatic cancer: a pilot trial demonstrating safety. Radiat Oncol. 2013 Mar 1;8:44. doi: 10.1186/1748-717X-8-44. PMID 23452509
- [Background] Koong AC, Le QT, Ho A, Fong B, Fisher G, Cho C, Ford J, Poen J, Gibbs IC, Mehta VK, Kee S, Trueblood W, Yang G, Bastidas JA. Phase I study of stereotactic radiosurgery in patients with locally advanced pancreatic cancer. Int J Radiat Oncol Biol Phys. 2004 Mar 15;58(4):1017-21. doi: 10.1016/j.ijrobp.2003.11.004. PMID 15001240
- [Background] Koong AC, Christofferson E, Le QT, Goodman KA, Ho A, Kuo T, Ford JM, Fisher GA, Greco R, Norton J, Yang GP. Phase II study to assess the efficacy of conventionally fractionated radiotherapy followed by a stereotactic radiosurgery boost in patients with locally advanced pancreatic cancer. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):320-3. doi: 10.1016/j.ijrobp.2005.07.002. PMID 16168826
- [Background] Schellenberg D, Kim J, Christman-Skieller C, Chun CL, Columbo LA, Ford JM, Fisher GA, Kunz PL, Van Dam J, Quon A, Desser TS, Norton J, Hsu A, Maxim PG, Xing L, Goodman KA, Chang DT, Koong AC. Single-fraction stereotactic body radiation therapy and sequential gemcitabine for the treatment of locally advanced pancreatic cancer. Int J Radiat Oncol Biol Phys. 2011 Sep 1;81(1):181-8. doi: 10.1016/j.ijrobp.2010.05.006. Epub 2011 May 5. PMID 21549517
- [Background] Bae SH, Kim MS, Cho CK, Kang JK, Lee SY, Lee KN, Lee DH, Han CJ, Yang KY, Kim SB. Predictor of severe gastroduodenal toxicity after stereotactic body radiotherapy for abdominopelvic malignancies. Int J Radiat Oncol Biol Phys. 2012 Nov 15;84(4):e469-74. doi: 10.1016/j.ijrobp.2012.06.005. PMID 23078899
- [Background] Bae SH, Kim MS, Kim SY, Jang WI, Cho CK, Yoo HJ, Kim KB, Lee DH, Han CJ, Yang KY, Kim SB. Severe intestinal toxicity after stereotactic ablative radiotherapy for abdominopelvic malignancies. Int J Colorectal Dis. 2013 Dec;28(12):1707-13. doi: 10.1007/s00384-013-1717-6. Epub 2013 Jun 18. PMID 23775098
- [Background] Chuong MD, Springett GM, Freilich JM, Park CK, Weber JM, Mellon EA, Hodul PJ, Malafa MP, Meredith KL, Hoffe SE, Shridhar R. Stereotactic body radiation therapy for locally advanced and borderline resectable pancreatic cancer is effective and well tolerated. Int J Radiat Oncol Biol Phys. 2013 Jul 1;86(3):516-22. doi: 10.1016/j.ijrobp.2013.02.022. Epub 2013 Apr 5. PMID 23562768
- [Background] Mahadevan A, Miksad R, Goldstein M, Sullivan R, Bullock A, Buchbinder E, Pleskow D, Sawhney M, Kent T, Vollmer C, Callery M. Induction gemcitabine and stereotactic body radiotherapy for locally advanced nonmetastatic pancreas cancer. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e615-22. doi: 10.1016/j.ijrobp.2011.04.045. Epub 2011 Jun 12. PMID 21658854
- [Background] Chang DT, Schellenberg D, Shen J, Kim J, Goodman KA, Fisher GA, Ford JM, Desser T, Quon A, Koong AC. Stereotactic radiotherapy for unresectable adenocarcinoma of the pancreas. Cancer. 2009 Feb 1;115(3):665-72. doi: 10.1002/cncr.24059. PMID 19117351
- [Background] Hoyer M, Roed H, Sengelov L, Traberg A, Ohlhuis L, Pedersen J, Nellemann H, Kiil Berthelsen A, Eberholst F, Engelholm SA, von der Maase H. Phase-II study on stereotactic radiotherapy of locally advanced pancreatic carcinoma. Radiother Oncol. 2005 Jul;76(1):48-53. doi: 10.1016/j.radonc.2004.12.022. PMID 15990186
- [Background] Didolkar MS, Coleman CW, Brenner MJ, Chu KU, Olexa N, Stanwyck E, Yu A, Neerchal N, Rabinowitz S. Image-guided stereotactic radiosurgery for locally advanced pancreatic adenocarcinoma results of first 85 patients. J Gastrointest Surg. 2010 Oct;14(10):1547-59. doi: 10.1007/s11605-010-1323-7. Epub 2010 Sep 14. PMID 20839073
- [Background] Mahadevan A, Jain S, Goldstein M, Miksad R, Pleskow D, Sawhney M, Brennan D, Callery M, Vollmer C. Stereotactic body radiotherapy and gemcitabine for locally advanced pancreatic cancer. Int J Radiat Oncol Biol Phys. 2010 Nov 1;78(3):735-42. doi: 10.1016/j.ijrobp.2009.08.046. Epub 2010 Feb 18. PMID 20171803
- [Background] Polistina F, Costantin G, Casamassima F, Francescon P, Guglielmi R, Panizzoni G, Febbraro A, Ambrosino G. Unresectable locally advanced pancreatic cancer: a multimodal treatment using neoadjuvant chemoradiotherapy (gemcitabine plus stereotactic radiosurgery) and subsequent surgical exploration. Ann Surg Oncol. 2010 Aug;17(8):2092-101. doi: 10.1245/s10434-010-1019-y. Epub 2010 Mar 12. PMID 20224860
- [Background] Rwigema JC, Parikh SD, Heron DE, Howell M, Zeh H, Moser AJ, Bahary N, Quinn A, Burton SA. Stereotactic body radiotherapy in the treatment of advanced adenocarcinoma of the pancreas. Am J Clin Oncol. 2011 Feb;34(1):63-9. doi: 10.1097/COC.0b013e3181d270b4. PMID 20308870
- [Background] Schellenberg D, Goodman KA, Lee F, Chang S, Kuo T, Ford JM, Fisher GA, Quon A, Desser TS, Norton J, Greco R, Yang GP, Koong AC. Gemcitabine chemotherapy and single-fraction stereotactic body radiotherapy for locally advanced pancreatic cancer. Int J Radiat Oncol Biol Phys. 2008 Nov 1;72(3):678-86. doi: 10.1016/j.ijrobp.2008.01.051. Epub 2008 Apr 18. PMID 18395362
- [Background] Goyal K, Einstein D, Ibarra RA, Yao M, Kunos C, Ellis R, Brindle J, Singh D, Hardacre J, Zhang Y, Fabians J, Funkhouser G, Machtay M, Sanabria JR. Stereotactic body radiation therapy for nonresectable tumors of the pancreas. J Surg Res. 2012 May 15;174(2):319-25. doi: 10.1016/j.jss.2011.07.044. Epub 2011 Sep 5. PMID 21937061
- [Background] Lominska CE, Unger K, Nasr NM, Haddad N, Gagnon G. Stereotactic body radiation therapy for reirradiation of localized adenocarcinoma of the pancreas. Radiat Oncol. 2012 May 18;7:74. doi: 10.1186/1748-717X-7-74. PMID 22607687
- [Background] Kavanagh BD, Schefter TE, Cardenes HR, Stieber VW, Raben D, Timmerman RD, McCarter MD, Burri S, Nedzi LA, Sawyer TE, Gaspar LE. Interim analysis of a prospective phase I/II trial of SBRT for liver metastases. Acta Oncol. 2006;45(7):848-55. doi: 10.1080/02841860600904870. PMID 16982549
- [Background] Rusthoven KE, Kavanagh BD, Cardenes H, Stieber VW, Burri SH, Feigenberg SJ, Chidel MA, Pugh TJ, Franklin W, Kane M, Gaspar LE, Schefter TE. Multi-institutional phase I/II trial of stereotactic body radiation therapy for liver metastases. J Clin Oncol. 2009 Apr 1;27(10):1572-8. doi: 10.1200/JCO.2008.19.6329. Epub 2009 Mar 2. PMID 19255321
- [Background] Kavanagh BD, Pan CC, Dawson LA, Das SK, Li XA, Ten Haken RK, Miften M. Radiation dose-volume effects in the stomach and small bowel. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S101-7. doi: 10.1016/j.ijrobp.2009.05.071. PMID 20171503
- [Derived] Qing S, Gu L, Zhang H. Phase I study of dose-escalated stereotactic body radiation therapy for locally advanced pancreatic head cancers: Initial clinical results. Cancer Med. 2021 Oct;10(19):6736-6743. doi: 10.1002/cam4.4214. Epub 2021 Aug 18. PMID 34405577
- [Derived] Qing SW, Ju XP, Cao YS, Zhang HJ. Dose escalation of Stereotactic Body Radiotherapy (SBRT) for locally advanced unresectable pancreatic cancer patients with CyberKnife: protocol of a phase I study. Radiat Oncol. 2017 Jan 9;12(1):6. doi: 10.1186/s13014-016-0760-1. PMID 28069017